CLINICAL TRIAL: NCT06940505
Title: Telemedicine Follow-up for Pre-malignant and Malignant Glottic Lesions: a Randomised Controlled Trial Study Protocol Comparing Care Close to Home Versus Standard of Care
Brief Title: Telemedicine Follow-Up for Early Laryngeal Cancer: a Randomized Controlled Trial Comparing Care Close to Home Versus Standard of Care
Acronym: Telemedicine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Isala (Other); Saxenburgh Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: M23.325004
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancers; Laryngeal Carcinoma
Keywords: head and neck cancer; follow-up; patient satisfaction; telemedicine; patient reported outcome measures; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Neoplasms; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine Group - Intervention (Experimental): Participants in the intervention group will receive follow-up care at a general hospital located nearby their residence. They will have a travel time reduction of ≥ 40%. During these visits, a general otolaryngologist will perform guideline-based follow-up evaluations, including high-definition laryngoscopy. The recorded endoscopic videos will be securely transferred and remotely evaluated by specialists at the Head and Neck Oncology Centre (HNOC) via Telemedicine. This collaborative model allows for specialist oversight without requiring the patient to travel long distances, aiming to maintain high standards of care while improving accessibility and convenience.
  Interventions: Other: Telemedicine Follow-up
- Control group (No Intervention): Participants in the control group (standard of care) will receive their follow-up care directly at the Head and Neck Oncology Centre (HNOC), in accordance with national guidelines. Follow-up visits will include in-person evaluations by a specialized head and neck oncologist, including high-definition laryngoscopy performed and interpreted on-site. This group represents the current standard practice for follow-up care in the Netherlands and serves as the control (long travel time) for evaluating patient satisfaction and safety in comparison to the Telemedicine model.

INTERVENTIONS:
Other: Telemedicine Follow-up — Oncological follow-up in a general hospital close to the patient, with aid of Telemedicine evaluation of the endoscopy video's by a Head and Neck surgeon in a specialised oncology centre
  Arms: Telemedicine Group - Intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether Telemedicine follow-up is a satisfactory and safe alternative to traditional follow-up care for patients treated for early glottic (vocal cord) cancer, particularly those who live far from a specialized head and neck oncology centre (HNOC).

The main questions it aims to answer are:

Is patient satisfaction with Telemedicine follow-up comparable to standard care?

Is the safety of Telemedicine follow-up (measured by recurrence rates, complications, and survival) comparable to in-person follow-up at an HNOC?

Researchers will compare patients receiving Telemedicine follow-up in a nearby hospital with standard in-person follow-up at the HNOC, to see if remote evaluation of endoscopic procedures can maintain patient satisfaction and safety outcomes.

Participants with a travel time of > 45 minutes from a HNOC will:

Be randomly assigned to either a Telemedicine follow-up group (in a nearby hospital, by a general ENT-surgeon) or a standard of care group

Undergo follow-up including HD-laryngoscopy, according to clinical guidelines

Have endoscopy videos evaluated remotely by specialists at the HNOC (= Telemedicine) (intervention group only)

Complete surveys including patient-reported outcomes and experience measures at baseline, 6 months, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent TOLS for early stage glottic squamous cell carcinoma (T1 or carcinoma-in-situ)
* a one-way travel time to the HNOC of ≥45 minutes (intervention group) or < 30 minutes (control group)
* within 2 years postoperatively
* can speak and write Dutch

Exclusion Criteria:

* Patients will be excluded if they continue to undergo follow-up for other (head and neck) cancers in the HNOC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 12 months
  Our primary outcomes are satisfaction with care and travel distance. Satisfaction is reported on a 0-10 numerical rating scale (NRS) and will be compared between study groups at baseline and 6 months and 12 months post-inclusion.
Patient satisfaction | 12 months
  Specific questions from the Consumer Quality Index (CQI) questionnaires are used for assessing patient satisfaction
Local and regional recurrence rate | 12 months
  Safety is measured by addressing local and regional recurrence rate
Postoperative complications after recurrence | 12 months
  Safety: postoperative complications after recurrence
Re-referral to the head and neck oncology center | 12 months
  Safety: re-referral rates to the oncology center
Disease specific and overall survival | 12 months
  Safety: survival

OTHER OUTCOMES:
HRQoL | 12 months
  In addition, the following outcome measures will be assessed: health related quality-of-life (HRQoL) using the ED-5D-5L questionnaire
Symptom burden | 12 months
  Using specific questions from the EORTC QLQ - H&N35 questionnaire
Fear of disease recurrence | 12 months
  Using the Cancer Worry scale
Traveling time and distance | 12 months
  Travel time in hours and minutes, distance in kilometres
Number of visits to the hospital | 12 months
  Amount of hospital visits

CONTACTS AND LOCATIONS:
Overall Officials: Boudewijn E.C. Plaat, MD, PhD, Principal Investigator — UMC Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Participants will not provide explicit consent for their data to be shared beyond the scope of the current study